CLINICAL TRIAL: NCT01516528
Title: Assessment of Comorbidities in Chronic Obstructive Pulmonary Disease (COPD) in European Symptomatic Subjects From Primary Care
Acronym: ACCESS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115058
Record Dates: First submitted 2012-01-12; First posted 2012-01-25 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; exacerbation; comorbidities; lung function; burden; chronic bronchitis; emphysema; prevalence; cardiovascular disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All: All subjects enrolled in the study
  Interventions: Procedure: Spirometry

INTERVENTIONS:
Procedure: Spirometry — Assessment of lung function by spirometry

SUMMARY:
This is a prospective, observational, non-drug interventional, non-randomized study to compare the rate of moderate-severe COPD exacerbations in patients of all Chronic Obstructive Pulmonary Disease (COPD) severities with and without cardiovascular diseases. A total study population of 3330 subjects will be recruited by general practitioners (GPs) and assessed over a 27 month time frame.

DETAILED DESCRIPTION:
COPD is a leading cause of morbidity and mortality worldwide. Comorbid diseases are an important factor in the prognosis and functional capabilities of COPD patients. There is a relationship between cardiac comorbidity and COPD exacerbation frequency within COPD patients. The main objective of this study is to compare the rate of moderate-severe COPD exacerbations in patients of all COPD severities with and without cardiovascular diseases. Secondary objectives will characterize the prevalence, severity and incidence over time of comorbidities and explore the relationships between comorbidities and rate of COPD exacerbations, force expiratory volume in 1 second (FEV1) decline and quality of life. This will be a prospective, observational, non-drug interventional, non-randomized study that will be carried out in up to 8 European countries. All patients will be enrolled by GP outpatient clinics and data will be collected over 4 visits (screening [-3 months], baseline, 12 months post baseline 24 months post baseline) and, additionally by 6 telephone calls (at 3, 6, 9, 15, 18 and 21 months post baseline). The study population will consist of 3330 evaluable patients with diagnosed COPD of any severity grade with and without comorbidities. Subjective and objective data on pre-defined comorbidities will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 40 years
* An established clinical history of COPD for a minimum of 12 months, of any severity.
* FEV1/FVC post-bronchodilator ratio < 0.70 (within the last 12 months, or confirmed at the screening visit [or 4 weeks after the screening visit if patient's COPD is not stable]).
* Current or ex-smokers with a smoking history of at least 10 pack-years
* A signed and dated written informed consent is obtained prior to participation

Exclusion Criteria:

* In the opinion of the investigator, there is a current primary diagnosis of asthma (patients with a primary diagnosis of COPD but who also have asthma may be included)
* A diagnosis of fibrosis or asbestosis
* Diagnosis of cancer - current or within the last 5 years (patients in remission for ≥ 5 years may be included). Patients diagnosed with cancer during the study will be withdrawn
* Diagnosis of clinically significant bronchiectasis
* Subjects who are concurrently participating in any clinical study or who have received any investigational drugs within 4 weeks of baseline, or who will start any during the study period.
* Unable to or unwilling to conform with the study requirements including completion of the health status questionnaires
* Females who are pregnant or lactating.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care outpatients who have a an established clinical history of COPD for a minimum of 12 months.
Sampling Method: Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2011-11-17; Primary Completion 2015-05-01 (Actual); Study Completion 2015-06-12 (Actual)

PRIMARY OUTCOMES:
Frequency of COPD Exacerbation | From 15 months pre-baseline to 24 months post-baseline.
  COPD exacerbations (moderate-severe severity), defined as a worsening of symptoms that require oral corticosteroids or antibiotics or hospitalization, or any combination of these.
Presence and severity of cardiovascular disease. | From 3 months pre-baseline to 24 months post-baseline.
  The presence and severity pre-defined cardiovascular diseases.

SECONDARY OUTCOMES:
Presence and severity of other comorbidities | Up to 24 months post baseline.
  The presence and severity of pre-defined comorbidities (depression/anxiety, diabetes with and without target organ disease, sleep apnoea syndrome, gastroesophageal reflux, hypercholesterolemia, osteoarthritis, osteoporosis, inflammatory bowel disease, peptic ulcer, other treated comorbidities) .
Spirometry | Up to 24 months post baseline.
  Post-bronchodilator FEV1 and forced vital capacity (FVC), FEV1/FVC ratio and FEV1 % of predicted.
Health status | Up to 24 months post baseline.
  As determined by COPD Assessment Test (CAT), EuroQOL Five Dimensions Questionnaire (EQ-5D), Hospital Anxiety Depression Scale (HADS) and Epworth Sleepiness Scale (ESS), Frequency Scale for the Symptoms of Gastro-oesophageal reflux disease (FSSG).
Dyspnoea | Up to 24 months post baseline.
  As determined by the modified Medical Research Council (mMRC) scale.
Number of Deaths | up to 24 months post baseline.
  Patients who die during the study, including the reason for death, where known.
Healthcare Utilisation | Up to 24 months post baseline.
  Number of unscheduled GP contacts and Hospitalisations
Blood Chemistry | Up to 24 months post baseline.
  Including glucose; Haemoglobin A1C (HbA1c); low density lipoprotein (LDL-c), High density lipoprotein (HDL-c), Total cholesterol; triglycerides, prohormone natriuretic peptide (pro-BNP); high-sensitivity C reactive protein (hs-CRP); protein; full blood count
Electrocardiogram | Up to 24 months post baseline.
  Assessment of normal or abnormal readings. Qualitative description and QT interval.
Bone fractures | Within 12 months prior to baseline and up to 24 months post baseline
  The number and location of bone fractures.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (200):
- GSK Investigational Site, Leuven, Belgium
- France (89):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Aumetz
  - GSK Investigational Site, Béziers
  - GSK Investigational Site, Blois
  - GSK Investigational Site, Bono
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Bouliac
  - GSK Investigational Site, Bourg-des-Comptes
  - GSK Investigational Site, Briollay
  - GSK Investigational Site, Carbon-Blanc
  - GSK Investigational Site, Carbonne
  - GSK Investigational Site, Chatou
  - GSK Investigational Site, Châtellerault
  - GSK Investigational Site, Cholet
  - GSK Investigational Site, Chollet
  - GSK Investigational Site, Couzeix
  - GSK Investigational Site, Cugnaux
  - GSK Investigational Site, Dinard
  - GSK Investigational Site, Donges
  - GSK Investigational Site, Franconville
  - GSK Investigational Site, Gémozac
  - GSK Investigational Site, Grandchamps
  - GSK Investigational Site, Haute-Goulaine
  - GSK Investigational Site, Houilles
  - GSK Investigational Site, La Baule-Escoublac
  - GSK Investigational Site, La Bouëxière
  - GSK Investigational Site, La Fôret Sur Sèvres
  - GSK Investigational Site, La Fresnais
  - GSK Investigational Site, La Jubaudière
  - GSK Investigational Site, La Montagne
  - GSK Investigational Site, La Riche
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, La Teste-de-Buch
  - GSK Investigational Site, La Varenne
  - GSK Investigational Site, Le Fousseret
  - GSK Investigational Site, Le Mesnil-en-Vallée
  - GSK Investigational Site, Les Ponts-de-Cé
  - GSK Investigational Site, Liffré
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Louvigné-de-Bais
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Martin-Église
  - GSK Investigational Site, Montreuil-Juigné
  - GSK Investigational Site, Montrevault
  - GSK Investigational Site, Mouliherne
  - GSK Investigational Site, Moulins-lès-Metz
  - GSK Investigational Site, Muret
  - GSK Investigational Site, Mûrs-Erigné
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nexon
  - GSK Investigational Site, Nieul-sur-Mer
  - GSK Investigational Site, Parçay-les-Pins
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Périgny
  - GSK Investigational Site, Pont-à-Mousson
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Royan
  - GSK Investigational Site, Saint-Aubin-des-Châteaux
  - GSK Investigational Site, Saint-Cyr-sur-Loire
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Étienne-de-Montluc
  - GSK Investigational Site, Saint-Georges-de-Montaigu
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Saint-Jouan-des-Guérets
  - GSK Investigational Site, Saint-Loubès
  - GSK Investigational Site, Saint-Max
  - GSK Investigational Site, Saint-Médard-en-Jalles
  - GSK Investigational Site, Saint-Orens-de-Gameville
  - GSK Investigational Site, Saint-Pierre-en-Val
  - GSK Investigational Site, Sarrebourg
  - GSK Investigational Site, Savonnières
  - GSK Investigational Site, Scorbé-Clairvaux
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Seysses
  - GSK Investigational Site, St-Malo
  - GSK Investigational Site, Thionville
  - GSK Investigational Site, Thouars
  - GSK Investigational Site, Tiercé
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vannes
  - GSK Investigational Site, Verzy
  - GSK Investigational Site, Vihiers
  - GSK Investigational Site, Villey-Saint-Étienne
  - GSK Investigational Site, Vitré
  - GSK Investigational Site, Vue
  - GSK Investigational Site, Witry-lès-Reims
  - GSK Investigational Site, Yerres
- Germany (38):
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Ettlingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Messkirch, Baden-Wurttemberg
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Bad Woerrishofen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Bensheim, Hesse
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Kelkheim, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Wardenburg, Lower Saxony
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Hagen, North Rhine-Westphalia
  - GSK Investigational Site, Harsewinkel, North Rhine-Westphalia
  - GSK Investigational Site, Rheine, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Ingelheim, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Nußbach, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Riesa, Saxony
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Zerbst, Saxony-Anhalt
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Reinfeld, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Netherlands (19):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Andijk
  - GSK Investigational Site, Beek en Donk
  - GSK Investigational Site, Deurne
  - GSK Investigational Site, Eersel
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Ermelo
  - GSK Investigational Site, Hoogwoud
  - GSK Investigational Site, Kloosterhaar
  - GSK Investigational Site, Lieshout
  - GSK Investigational Site, Musselkanaal
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Soerendonk
  - GSK Investigational Site, Spijkenisse
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Voerendaal
  - GSK Investigational Site, Wildervank
  - GSK Investigational Site, Zaandam
  - GSK Investigational Site, Zwijndrecht
- Poland (23):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Domaradz
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Jasło
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Libiąż
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Mielec
  - GSK Investigational Site, Oświęcim
  - GSK Investigational Site, Puławy
  - GSK Investigational Site, Radom
  - GSK Investigational Site, Radziszów
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zabrze
  - GSK Investigational Site, Zgierz
  - GSK Investigational Site, Zgłobień
- Spain (30):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Algeciras
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barakaldo
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benidor / Alicante
  - GSK Investigational Site, Canet de Mar - Barcelona
  - GSK Investigational Site, Colloto - Oviedo
  - GSK Investigational Site, Cornellá de Llobregat-Barcelona
  - GSK Investigational Site, Culleredo - La Coruña
  - GSK Investigational Site, El Puerto de Santa María-Cádiz
  - GSK Investigational Site, Fuenlabrada / Madrid
  - GSK Investigational Site, Gijón
  - GSK Investigational Site, Gijón. Asturias.
  - GSK Investigational Site, Güeñes - Vizcaya
  - GSK Investigational Site, Hostalric - Gerona
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Les Franqueses Del Vallés - Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Mataró. Barcelona.
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Peralada( Girona)
  - GSK Investigational Site, Petrer/Alicante
  - GSK Investigational Site, Portugalete - Vizcaya
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, Santa Coloma de Gramanet - Barcelona
  - GSK Investigational Site, Valencia